CLINICAL TRIAL: NCT00348426
Title: Clinical Manifestations of Botulism Outbreak in Northern Thailand: A Case Series of Botulism Treated With Botulinum Anti-Toxin.
Brief Title: Botulism Outbreak in Thailand (Episode II)
Status: Completed | Type: Observational
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Collaborators: Rajavithi Biomolecular Research Center (Other)
Other Study IDs: RVH_CER_002
Record Dates: First submitted 2006-07-02; First posted 2006-07-04 (Estimated); Last update posted 2006-11-08 (Estimated); Status verified 2006-11

CONDITIONS: Botulism
Keywords: Food Borne Botulism
MeSH Terms: conditions — Botulism | interventions — Botulinum Antitoxin

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: Botulinum AntiToxin
Procedure: neuro-electrophysiologic study, repetitive nerve stimulation
Procedure: : Protocol early weaning ventilator after recovery of repetitive nerve stimulation and stable negative inspiratory pressure

SUMMARY:
A second botulism outbreak in Northern Thailand was reported in 2006. 192 people were exposed to raw meat and the gut of deer, 83 suffered from diarrhea. Of these 5 developed respiratory failure, 1 impending respiratory failure.

We analysed the clinical findings and electrophysiologic findings in this second episode of large botulism outbreak in northern Thailand.

DETAILED DESCRIPTION:
PRELIMINARY REPORT Northern Thailand's big botulism outbreak occurred again on 30 June 14, 2006, [16.00pm] affecting 83 from 192 people who exposed to raw dear meat and gut [1 night preserved with ice pack of whole body of dear before disection and distribution ]. Of these, 3 developed respiratory failure, 1 developed impending respiratory failure, 83 of 192 whom developed fatique and diarrhea after ingestion of raw dear meat and gut on 26-30 June 2006. 3 patients were refered to 2 high facility hospitals for severe respiratory failure. Physical examination of 3 patients in ICU of Chiang Kum general hospital revealed ptosis [3/3] mild ophthalmoparesis [2/3] Proximal muscle weakness [2/3] abdominal paradoxical respiration [3/3] pupil dilate [1/3] and negative inspiratory pressure [NIP] less than 15 mmHg [3/3] were observed. Neurological electrophysiologic study of 2 patients revealed low amplitude compound muscle action potential [CMAP] of Abductor digiti minimi [ADM] muscle with decrement response after repetitive stimulation with low frequency [3Hz], increment response of ADM muscle after stimulation with high frequency [10Hz, 20Hz, and 30Hz.].The electrophysiologic findings support diagnosis of presynaptic neuromuscular dysfunction with respiratory failure, Botulism is most likely diagnosis. After treated with botulinum antitoxin [on July,1 ,2006 [mixed-type botulinum antitoxin --donated from Japan at Nan Hospital's botulisum outbreak on March 14,2006], 3 patients in ICU showed improvement of over all clinical outcomes. Active survey by Ministry of Public Health of Thailand and CDC-USA to identify the high risk patient who may develop respiratory failure , and immunologucal vs microbiological diagnosis were performed. This outbreak may be the second hit of botulisum in the northern Thailand but less amount of severe cases was observed.

ELIGIBILITY:
Inclusion Criteria:

* Ate the deer meat and/or the gut from Chiang Kum district, after June 26,2006
* Clinical botulism or respiratory failure who need ventilator assistance
* The staff of referring hospital willing to participate in the Thai Botulism study group

Exclusion Criteria:

• Patients who did not eat deer meat and or the gut from Chiang Kum district

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2006-06; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Subsai Kongsaengdao, M.D., Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Chiang Kum Hospital, Payao, Payao, Thailand

REFERENCES:
- [Background] World Health Organization .Botulism in Thailand: Epidemic and Pandemic Alert and Response (EPR). (Accessed March 22, 2006, at http://www.who.int/csr/don/2005_12_22/en/)
- [Background] P Wongwatcharapaiboon, L Thaikruea, and K Ungchusak et. al. Foodborne Botulism Associated With Home-Canned Bamboo Shoots,Thailand, 1998. ). (Accessed March 22, 2006, at http://www.cdc.gov/mmwr/preview/mmwrhtml/mm4821a1.htm)
- [Background] Swaddiwudhipong W, Wongwatcharapaiboon P. Foodborne botulism outbreaks following consumption of home-canned bamboo shoots in Northern Thailand. J Med Assoc Thai. 2000 Sep;83(9):1021-5. PMID 11075968
- [Background] Fernandez PS, Peck MW. A predictive model that describes the effect of prolonged heating at 70 to 90 degrees C and subsequent incubation at refrigeration temperatures on growth from spores and toxigenesis by nonproteolytic Clostridium botulinum in the presence of lysozyme. Appl Environ Microbiol. 1999 Aug;65(8):3449-57. doi: 10.1128/AEM.65.8.3449-3457.1999. PMID 10427033
- [Background] Jones RG, Corbel MJ, Sesardic D. A review of WHO International Standards for botulinum antitoxins. Biologicals. 2006 Sep;34(3):223-6. doi: 10.1016/j.biologicals.2005.11.009. Epub 2006 Feb 20. PMID 16490362
- [Background] Sobel J, Tucker N, Sulka A, McLaughlin J, Maslanka S. Foodborne botulism in the United States, 1990-2000. Emerg Infect Dis. 2004 Sep;10(9):1606-11. doi: 10.3201/eid1009.030745. PMID 15498163
- [Background] Boyadjiev I, Leone M, Garnier F, Thomachot L, Martin C. [A case of type A botulism]. Ann Fr Anesth Reanim. 2005 Nov-Dec;24(11-12):1397-9. doi: 10.1016/j.annfar.2005.06.002. Epub 2005 Oct 26. French. PMID 16256299
- [Background] Sobel J. Botulism. Clin Infect Dis. 2005 Oct 15;41(8):1167-73. doi: 10.1086/444507. Epub 2005 Aug 29. PMID 16163636
- [Background] Agarwal AK, Goel A, Kohli A, Rohtagi A, Kumar R. Food-borne botulism. J Assoc Physicians India. 2004 Aug;52:677-8. No abstract available. PMID 15847370
- [Background] Kongsaengdao S, Samintarapanya K, Rusmeechan S, Wongsa A, Pothirat C, Permpikul C, Pongpakdee S, Puavilai W, Kateruttanakul P, Phengtham U, Panjapornpon K, Janma J, Piyavechviratana K, Sithinamsuwan P, Deesomchok A, Tongyoo S, Vilaichone W, Boonyapisit K, Mayotarn S, Piya-Isragul B, Rattanaphon A, Intalapaporn P, Dusitanond P, Harnsomburana P, Laowittawas W, Chairangsaris P, Suwantamee J, Wongmek W, Ratanarat R, Poompichate A, Panyadilok H, Sutcharitchan N, Chuesuwan A, Oranrigsupau P, Sutthapas C, Tanprawate S, Lorsuwansiri J, Phattana N; Thai Botulism Study Group. An outbreak of botulism in Thailand: clinical manifestations and management of severe respiratory failure. Clin Infect Dis. 2006 Nov 15;43(10):1247-56. doi: 10.1086/508176. Epub 2006 Oct 16. PMID 17051488